CLINICAL TRIAL: NCT04965168
Title: Evaluation of Corneal Endothelium Following Phacoemulsification in Diabetic and Non-diabetic Patients With Pseudoexfoliation Syndrome by Specular Microscopy
Brief Title: Corneal Endothelium Evaluation After Phacoemulsification in Diabetec and Non-diabetic Patients With Pseudoexfoliation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Heba Radi AttaAllah, Associate Professor of Ophthalmology, Minia University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 691:11/2020
Record Dates: First submitted 2021-07-07; First posted 2021-07-16 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Pseudoexfoliation
Keywords: DM; phacoemulsification; endothelial cell density

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- controls (Active Comparator): phacoemulsification and IOL implantation
  Interventions: Procedure: phacoemulsification of the lens
- diabetic without pseudoexfoliation (Active Comparator): phacoemulsification and IOL implantation
  Interventions: Procedure: phacoemulsification of the lens
- non-diabetic with pseudoexfoliation (Active Comparator): phacoemulsification and IOL implantation
  Interventions: Procedure: phacoemulsification of the lens
- diabetic with pseudoexfoliation (Active Comparator): phacoemulsification and IOL implantation
  Interventions: Procedure: phacoemulsification of the lens

INTERVENTIONS:
Procedure: phacoemulsification of the lens — all patients underwent phacoemulsification and IOL implantation for immature cataract extraction

SUMMARY:
Our study is a comparative study, that was conducted to evaluate the corneal endothelial cells changes and central corneal thickness after uncomplicated phacoemulsification and intra ocular lens (IOL) implantation in normal controls, in non-diabetic and diabetic patients with PEX, and in patients with PEX only using specular microscopy.

DETAILED DESCRIPTION:
Our study is a comparative study that included 4 groups (controls, patients with PEX, non-diabetic patients with PEX, diabetic patients with PEX) to evaluate the corneal endothelial cells changes and central corneal thickness after uncomplicated phacoemulsification and intra ocular lens (IOL) implantation using specular microscopy, over a 6 months follow up period.

ELIGIBILITY:
Inclusion Criteria:

* Senile cataract with age between 50 to 70 years
* Clear cornea with no zonuler dehiscence
* Lens opacity classification system III (LOCS III), with grade 2-3 nuclear cataract with any additional cortical (C) and posterior sub capsular (P)

Exclusion Criteria:

* Uncontrolled DM in diabetic groups
* Presence of autoimmune diseases
* Patients with glaucoma
* Corneal guttata
* Zonular dehiscence
* Rupture posterior capsule during cataract surgery

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-10-12 (Actual); Study Completion 2021-10-16 (Actual)

PRIMARY OUTCOMES:
endothelial cell density | 6 months
  number of endothelial cells
Percentage of hexagonal cells | 6 months
  indicator of healthy endothelial cells
coefficient of variation (CV) | 6 months
  indicator of the uniformity of the size of endothelial cells
Central corneal thickness | 6 months
  measurement of the distance between the epithelium and endothelium at the central cornea

CONTACTS AND LOCATIONS:
Overall Officials: Heba R AttaAllah, MD, Principal Investigator — Faculty of Medicine, Minia University
Locations (1):
- Ophthalmology department/ Minia University Hospital/Minia University, Minya, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Storr-Paulsen A, Singh A, Jeppesen H, Norregaard JC, Thulesen J. Corneal endothelial morphology and central thickness in patients with type II diabetes mellitus. Acta Ophthalmol. 2014 Mar;92(2):158-60. doi: 10.1111/aos.12064. Epub 2013 Feb 7. PMID 23387877
- [Background] Fernandez-Munoz E, Zamora-Ortiz R, Gonzalez-Salinas R. Endothelial cell density changes in diabetic and nondiabetic eyes undergoing phacoemulsification employing phaco-chop technique. Int Ophthalmol. 2019 Aug;39(8):1735-1741. doi: 10.1007/s10792-018-0995-y. Epub 2018 Jul 28. PMID 30056522
- [Background] Oltulu R, Satirtav G, Kayitmazbatir ET, Bitirgen G, Ozkagnici A, Karaibrahimoglu A. Characteristics of the cornea in patients with pseudoexfoliation syndrome. Arq Bras Oftalmol. 2015 Nov-Dec;78(6):348-51. doi: 10.5935/0004-2749.20150092. PMID 26677035
- [Background] Aoki T, Kitazawa K, Inatomi T, Kusada N, Horiuchi N, Takeda K, Yokoi N, Kinoshita S, Sotozono C. Publisher Correction: Risk Factors for Corneal Endothelial Cell Loss in Patients with Pseudoexfoliation Syndrome. Sci Rep. 2020 May 26;10(1):8800. doi: 10.1038/s41598-020-66089-4. PMID 32451432
- [Background] Quiroga L, Lansingh VC, Samudio M, Pena FY, Carter MJ. Characteristics of the corneal endothelium and pseudoexfoliation syndrome in patients with senile cataract. Clin Exp Ophthalmol. 2010 Jul;38(5):449-55. doi: 10.1111/j.1442-9071.2010.02313.x. Epub 2010 Apr 28. PMID 20456430
- [Derived] Mahmoud MSE, Omar IAN, AttaAllah HR. Evaluation of the corneal thickness and endothelial changes following uncomplicated phacoemulsification in diabetic and non-diabetic patients with pseudo-exfoliation syndrome by specular microscopy. Int Ophthalmol. 2023 Dec;43(12):4773-4780. doi: 10.1007/s10792-023-02877-x. Epub 2023 Sep 18. PMID 37721703